CLINICAL TRIAL: NCT03866798
Title: Post-Marketing Study to Evaluate the Efficacy and Safety of PANZYGA in Pediatric Patients With Chronic Immune Thrombocytopenia (ITP)
Brief Title: Study to Evaluate the Efficacy and Safety of PANZYGA in Pediatric Patients With Chronic Immune Thrombocytopenia (ITP)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: FDA released Octapharma from the pediatric post marketing requirement.
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGAM-10
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Chronic Immune Thrombocytopenia
MeSH Terms: interventions — Panzyga

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Panzyga (Experimental): Panzyga
  Interventions: Biological: Panzyga

INTERVENTIONS:
Biological: Panzyga — Immune Globulin, intravenous, human-ifas

SUMMARY:
This is a prospective, open-label, single-arm, multicenter, Phase 4 study evaluating the efficacy and safety of PANZYGA in pediatric patients with chronic ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males aged from ≥1 year to <18 years old
2. Confirmed diagnosis of Chronic Immune Thrombocytopenia (ITP) according to American Society of Hematology (ASH) 2019 guidelines
3. Platelets count <30x10^9/L at the Baseline Visit
4. Voluntarily given written informed consent (provided by patient's parent or legal guardian) and assent (provided by patient [if age-appropriate per IRB (Institutional Review Board) requirements])
5. Sexually active females who have been using at least 1 acceptable form of birth control for a minimum of 30 days (or a minimum of 3 months for hormonal contraceptives) prior to the Screening visit and must agree to use at least 1 acceptable method of contraception throughout the study and for 30 days after the last dose of PANZYGA. Acceptable methods of birth control for this study include: intrauterine device (IUD), hormonal contraception, male or female condom, spermicide gel, diaphragm, sponge, or cervical cap. For non-sexually active females who have begun menstruating, abstinence is considered an acceptable method of birth control.
6. Parent or legal guardian must agree and be willing to assist the participant attend study visits, and to follow all protocol requirements and instructions of the study doctor

Exclusion Criteria:

1. Thrombocytopenia secondary to other diseases (such as Acquired Immunodeficiency Syndrome [AIDS] or systemic lupus erythematosus [SLE]), drug-related thrombocytopenia, or congenital thrombocytopenia
2. Administration of intravenous immunoglobulin (IGIV) or anti-D immunoglobulin within 3 weeks (+/- 3 days) before enrollment
3. Administration of thrombopoietin receptor agonists when the dose has NOT been stable within 3 weeks before enrollment and a dosage change is planned before Day 32
4. Administration of oral immunosuppressants when the dose has NOT been stable during the preceding 2 months (2 weeks for long-term corticosteroid therapy) and a dosage change is planned before Day 32 (Note: topical agents and inhaled corticosteroid therapy use is permitted)
5. Administration of long-term anti-prolific agents or attenuated androgen therapy when the dose has NOT been stable during the preceding 2 months and a dosage change is planned before Day 32
6. Nonresponsive to previous treatment with IGIV or anti-D immunoglobulin
7. Evidence of an active major bleeding episode at Screening
8. Splenectomy in the previous 3 months or planned splenectomy throughout the study period
9. Evans syndrome (experiencing active disease with 2 out of 3 of the following: autoimmune thrombocytopenia, autoimmune hemolytic anemia, and/or autoimmune neutropenia)
10. Known or suspected human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) infections
11. Emergency surgery in the previous 4 weeks
12. Severe liver and/or kidney disease (alanine aminotransferase [ALT] >3x upper limit of normal (ULN), aspartate aminotransferase [AST] >3x upper limit of normal (ULN), and/or creatinine >120 µmol/L)
13. History of severe hypersensitivity to blood or plasma derived products, or any component of the PANZYGA
14. Known immunoglobulin A (IgA) deficiency and antibodies against IgA
15. History of, or suspected alcohol or drug abuse in the previous year
16. Females who are pregnant or nursing
17. Unable or unwilling to comply with the study protocol
18. Receipt of any other investigational medicinal product within 3 months before study entry
19. Risk factors* for thromboembolic events in whom the risks outweigh the potential benefit of PANZYGA treatment.
20. Any other condition(s), that in the Investigator's opinion, make it undesirable for the patient to participate in the study or may interfere with protocol compliance.

    * Risk factors include, but are not limited to: obesity, advanced age, hypertension, diabetes, a history of atherosclerosis/vascular disease or thrombotic events, hyperlipidemia, multiple cardiovascular risk factors, acquired or inherited thrombophilic disorders, prolonged periods of immobilization, severe hypovolemia, central venous catheterization, active malignancy and/or known or suspected hyperviscosity.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Octapharma Research Site, Sacramento, California
  - Octapharma Research Site, Minneapolis, Minnesota
  - Octapharma Research Site, Rochester, Minnesota
  - Octapharma Research Site, Columbus, Ohio
  - Octapharma Research Site, Toledo, Ohio
  - Octapharma Research Site, Philadelphia, Pennsylvania
  - Octapharma Research Site, Providence, Rhode Island
  - Octapharma Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six subjects aged ≥1 year to <18 years were recruited between 21-Jan-2020 and 19-Sep-2023. The subjects were enrolled at five research sites across the United States, with a total of eight research sites activated in the study.
Period: Overall Study
Arm/Group | Panzyga
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Panzyga
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Platelet Count Increase
Description: Number of subjects with an increase in platelet count at least once to ≥50 × 10^9/L within 7 days after the first infusion, i.e., by Day 8 (increase must have occurred at least once on any day up to and including Day 8).
Time Frame: 8 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Panzyga
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Days to Reach Platelet Count of at Least 50x10^9/L
Description: Number of days for subjects to reach Platelet Count of at least 50x10^9/L after infusion
Time Frame: Through study completion, up to 37 days
Measure: Count of Participants; unit: Participants
Arm/Group | Panzyga
Number analyzed (Participants) | 6
Participants
  2 days | 3
  3 days | 1
  Did not reach Platelet Count of at least 50x10^9/L | 2

3. Secondary Outcome: Duration of Platelet Response
Description: Number of days the platelet count remains above at least 50x10^9/L
Time Frame: Through study completion, up to 37 days
Measure: Count of Participants; unit: Participants
Arm/Group | Panzyga
Number analyzed (Participants) | 6
Participants
  6 days | 1
  7 days | 1
  33 days | 1
  34 days | 1
  Did not reach Platelet Count of at least 50x10^9/L | 2

4. Secondary Outcome: Maximum Platelet Count
Description: Maximum platelet count (10^9/L) for each subjects
Time Frame: Through study completion, up to 37 days
Measure: Count of Participants; unit: Participants
Arm/Group | Panzyga
Number analyzed (Participants) | 6
Participants
  99 (10^9/L) | 1
  11 (10^9/L) | 1
  516 (10^9/L) | 1
  386 (10^9/L) | 1
  204 (10^9/L) | 1
  30 (10^9/L) | 1

ADVERSE EVENTS:
Time Frame: 3 years, 9 months
Arm/Group | Panzyga
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panzyga (N=6)
Headache (Nervous system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mouth haemorrhade (Gastrointestinal disorders) | 1 (2)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT03866798/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT03866798/SAP_001.pdf